CLINICAL TRIAL: NCT03808883
Title: Understanding and Reducing Health Disparities Faced by Transgender and Gender Non-conforming (TGNC) Individuals in Cleveland Through TGNC-Directed Advocacy
Brief Title: TRANSLATE: Transgender and Gender Nonconforming Individuals' Access to Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: LGBT Community Center of Greater Cleveland (Other); MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-2018-2194
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Gender Identity
Keywords: Barriers to Healthcare Access; Participatory Action Research; Cultural Competency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGNC Cohort (Experimental): The Translate Study developed a cohort of transgender and gender non-conforming individuals (referred to here as TGNC cohort) and held three facilitated dialogue sessions with healthcare providers and staff (referred to here as healthcare participants). The overall goal of the Translate Study was to improve quality of life by reducing health disparities suffered by transgender and gender nonconforming (TGNC) individuals and by increasing their access to and use of primary health care.
  Interventions: Behavioral: TGNC Directed Advocacy Meetings; Behavioral: Facilitated Dialogues between TGNC Cohort and Healthcare Participants
- Healthcare Participants (Experimental): The Translate Study held three facilitated dialogue sessions between the TGNC Cohort and a group of healthcare participants, identified as physicians, nurse practitioners, registered nurses, students, physician assistants, and non-provider staff positions. Non-providers included healthcare administrative positions, rehabilitation, and vocational services.
  Interventions: Behavioral: Facilitated Dialogues between TGNC Cohort and Healthcare Participants

INTERVENTIONS:
Behavioral: TGNC Directed Advocacy Meetings — Series of 18 meetings with TGNC cohort, including 3 facilitated dialogues with the healthcare participants, to articulate barriers to access and to enter into dialogue with medical providers and staff.
  Arms: TGNC Cohort
Behavioral: Facilitated Dialogues between TGNC Cohort and Healthcare Participants — Healthcare Participants attend a facilitated dialogue with the TGNC cohort. 3 total facilitated dialogues were held, but each healthcare participant attends only 1 session.

SUMMARY:
Transgender and gender nonconforming (TGNC) individuals face a number of health disparities, many of which can be tied to a lack of access to or use of primary care. Stigma and misunderstanding make simple doctor's visits into ordeals only worth enduring for the most serious of problems. This project addresses those issues by enlisting TGNC people as experts on their own experience. TGNC individuals will form a year-long cohort that will form the basis for this research. Collectively, they will define the scope of challenges faced when seeking healthcare, what medical advocacy training they desire, and how to address groups of healthcare providers and staff. Healthcare providers, including MDs, nurses, and Physicians Assistants (PAs), will attend two facilitated sessions with the TGNC cohort to meet as peers with knowledge exchanged in both directions. Similar meetings will occur with clinic staff, as TGNC individuals have expressed how stigma begins from the moment they call a medical office. Our hypothesis is that when TGNC individuals are given the tools to navigate the healthcare system and the ability to speak with medical professionals as peers, rather than patients, through a participatory action research design they will be better able to access appropriate care through increased confidence and mutual support. The complementary hypothesis for medical providers is that direct interaction with a variety of TGNC individuals who articulate their needs will decrease stigma and increase comfort when treating TGNC people as patients. As a partnership between academic, medical, and community institutions, this project has the potential to directly impact the lives of TGNC individuals who participate and indirectly impact others served by the LGBT Center. This proposal works on three levels: 1) at the academic level - an assessment of participatory action research as an intervention to decrease health disparities, 2) at the individual level - the potential for individuals to increase personal knowledge and skills, and 3) at the institutional level - as actors within the TGNC community develop relationships with individual healthcare providers, medical clinics and activist groups and community partners and educational institutions are concurrently forming networks that will have positive, although probably more diffuse, impact on TGNC individuals as these institutions come together to support TGNC health care.

DETAILED DESCRIPTION:
RESEARCH QUESTION: Do interactive dialogues between trans and gender nonconforming (TGNC) - trained in health literacy and advocacy - and healthcare providers and staff seeking cultural competency around TGNC primary care result in 1) more confidence on the part of TGNC in navigating the healthcare system, 2) more confidence on the part of providers in responding to the needs of TGNC patients, (sub question - is there a measurable difference between types of providers' responses to trainings, i.e., medical doctors compared to nurse practitioners) 3) person-to-person networks between the two populations resulting in ongoing, sustainable dialogue, 4) TGNC individuals prepared to train other TGNC in a peer-to-peer role to act as advocates on behalf of the TGNC population within the healthcare system, all of which ultimately result in increased access to and use of primary care services and reduce the health disparities faced by TGNC individuals? SIGNIFICANCE: The LGBTQ+ community has historically acted on its own behalf out of necessity, including for the push to remove homosexuality as a mental disorder from the The Diagnostic and Statistical Manual of Mental Disorders (DSM) and reframing the HIV/AIDS conversation and demanding research. Our project, driven by TGNC people's interests and advocacy, falls within this tradition of advocacy from inside the community. Our project aims to improve quality of life by addressing health disparities faced by TGNC individuals and by developing a self-sustained space to teach self-advocacy skills to navigate the healthcare system. The LGBT Community Center of Greater Cleveland (The LGBT Center) is in the process of hiring a new Youth Program Coordinator who will be responsible for the project management of this program. The ideal candidate will bring both professional and personal experience of working within the TGNC community and an interest in research. "TRANS in the CLE Conference," convened in October of 2017, had more than 130 attendees, 26 presenters, and 15 workshops. The LGBT Center regularly hosts the Queer Youth Initiative, serving an average of 100 people a month between the ages of 11 and 20. A majority of those individuals identify as transgender, non-binary, or gender nonconforming. This demonstrates both the significant presence of TGNC individuals in Cleveland and the LGBT Center's ability to reach this population.

INNOVATION: This project places TGNC community members and The LGBT Center in position to lead the direction of the research project, to gain research and health advocacy skills themselves, and the ability to form a cohort that will continue to operate beyond this pilot project. In Cleveland, TGNC affirming services are available at the Pride Network at MetroHealth, Cleveland Clinic's Center for LGBT Care, and University Hospital's navigator program. ECHO community partners receive technical assistance from experts in the field, but these are not necessarily informed by TGNC community input. Almost no other academic program is asking TGNC people what issues to prioritize, and no other program in the Cleveland area, to our knowledge. TGNC individuals are often research subjects and not recognized as experts themselves. Alpert's online survey asks LGBTQ+ individuals what they feel doctors should say and do, but the interaction is still mediated through an academic expert. The intervention closest to what is proposed is the Transgender Law's "Organizing for Transgender Healthcare: A Guide for Community Clinic Organizing and Activism", which defines transgender health care as "culturally appropriate primary health care, including access to sex-specific and transition-related procedures". In a case study in Los Angeles, a group of trans men formed an advocacy group (C3) that engaged with two community clinics to improve the clinics' cultural competency, medical forms, outreach materials, protocols for accessing hormones, and the referral process. This project is being proposed by cisgender women but is designed to be driven by TGNC individuals as partners and advocates navigating the healthcare system. In comparison to the model of C3 in Los Angeles, this project is innovative in that it calls for a sustained dialogue between the TGNC cohort and the health care providers and reaches a cross-section of practitioners from clinics that provide primary care.

METHODS: Over the course of the grant year, each step of the project is divided into three month portions. The first quarter will be dedicated to recruiting and forming a cohort of TGNC individuals, drawn mostly from the LGBT Center's extensive contact lists and centrality within the TGNC population. The investigators plan on recruiting 20 individuals to ensure the study meets the minimum retention of 12 subjects throughout the study needed for qualitative saturation, and individuals between 14-18 years of age will be able to participate with guardian permission. Interested individuals will fill out applications to identify their interests and ability to commit to the project and will allow us to create a cohort that reflects the diversity of the TGNC community in Cuyahoga County, including gender identity, types of gender-affirmative care required (including whether or not someone is considering, in the process of, or completed physical transition), racial and ethnic identity, age (over 14), and socio-economic class. Upon accepting the invitation to participate, each member of the cohort will complete a pretest that will elicit data on their experiences in the healthcare system, their knowledge of basic and transgender-specific medical terminology, their familiarity with healthcare providers in Cuyahoga County, and the likelihood of seeking care under a number of conditions (acute, chronic, moderate, severe). The investigators expect this to take one month. The following two months will consist of meeting as a cohort twice a month. The first two meetings will be dedicated to understanding the group's collective experiences with health care, what they would like to see change, and what strategies can be used to accomplish those ends. The investigators recognize that TGNC people come from a variety of backgrounds and each will bring their own strengths, networks, and perspectives to the table which will allow us to make full use of the indigenous expertise of the group. In consultation with the Nursing School of CWRU, the investigators will develop a health literacy training that meets the expressed needs of the cohort and Jesse Honsky will present it during the 3rd meeting. The goal here is not to provide all possible health education but rather to arm the cohort with the skills and language to empower them to act as advocates on their own behalf when navigating the healthcare system. The final meeting (the 4th) in this first quarter will be with a trained facilitator (Shemariah Arki) who will, under the direction of the TGNC cohort, plan a series of three interactive dialogues between the TGNC cohort and the healthcare providers. By meeting with the TGNC cohort first, without the healthcare providers, the TGNC cohort will have the opportunity to ensure the dialogues are designed to meet their objectives. Individual healthcare practitioners and medical staff will be recruited during the first quarter from the aforementioned clinics. The investigators will recruit at least twelve providers and twelve staff members. In the second quarter, the investigators will conduct a pretest that will collect data on attitudes towards TGNC individuals, TGNC-specific healthcare concerns, depth and breadth of referral networks for TGNC providers. Once the healthcare provider group is solidified, the LGBT Center will host three evening meetings (once per month) with the trained facilitator wherein TGNC individuals lead a conversation about what they see as barriers to their care, how they would like to be treated, and what they want healthcare providers to know about them as people. The first two meetings will be with healthcare practitioners and the final meeting will be medical staff so that the meetings can be more specific and without the interference of power dynamics within the provider groups. During this second quarter, the TGNC cohort will continue to meet on its own once a month to debrief from meetings, respond to what they have learned so far, and possibly refine the strategies for future meetings with healthcare providers as the series goes forward. At the end of the three months of dialogue, each participant, from both the TGNC cohort and healthcare provider, will be given a post-test to measure changes in attitude, practice, and knowledge. Participants will also have the opportunity to engage in a reflective interview.

The third quarter will diverge onto two different paths: the LGBT Center project coordinator will continue to engage with the cohort as they shift into the role of peer educators and advocates with other members of the TGNC community that interact at the LGBT Center. Luminais will conduct follow-up interviews with any TGNC cohort member that notifies the researchers that they have sought medical care and with any healthcare provider that notifies the researchers that they have had a clinical interaction with a TGNC individual. The investigators will not be seeking any protected medical information or the identity of patients, in the case of healthcare providers, but rather a discussion of the ease or difficulty in communication, levels of comfort, and comparison with other interactions in general.

Throughout the process, both Luminais and the LGBT Center coordinator will be engaged in participant observation and keep detailed field notes on all the meetings. All interviews will be transcribed; interviews and field notes will be coded with a priori codes derived from the literature on reducing health disparities and TGNC-specific health care by a research assistant. Pre- and post-tests will be analyzed to determine the success of facilitated dialogue in improving confidence and knowledge by both the TGNC cohort and the healthcare providers, and depending on sample size, the investigators will determine if there are any statistically significant changes. This analysis and write up will encompass the last quarter of the project.

ELIGIBILITY:
TGNC Inclusion Criteria:

* self-identify as transgender or gender nonconforming
* fluent English speaker
* above the age of 14 years old

TGNC Exclusion Criteria:

* non-fluent English speaker
* below the age of 14 years old
* does not identify as transgender or gender nonconforming

Healthcare Participants Inclusion Criteria:

* Currently employed as a medical provider or medical staff
* At least 18 years old
* fluent English speaker

Healthcare Participants Exclusion Criteria:

* Not currently employed as a medical provider or medical staff
* non-fluent English speaker
* below the age of 18 years old

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — TGNC cohort must self-identify as transgender or gender nonconforming
Enrollment: 49 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Flannery, PhD, Study Chair — Director, Begun Center for Violence Prevention Research and Education; Jack, Joseph and Morton Mandel School of Applied Social Sciences
Locations (1):
- LGBT Community Center of Greater Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TGNC Cohort: Transgender and gender non-conforming (TGNC) identifying individuals.
  TGNC Directed Advocacy Meetings: Series of 18 community meetings with TGNC individuals, 3 of which were facilitated dialogues with health professionals to articulate barriers to access and to enter into dialogue with medical providers and staff.
- Healthcare Participants: Healthcare Providers and staff who participated in a facilitated dialogue with the TGNC Cohort. The Translate Study held three facilitated dialogue sessions with both the TGNC Cohort and Healthcare Participants, identified as physicians, nurse practitioners, registered nurses, students, physician assistants, and non-provider staff positions. Each Healthcare Participant only attended one of the three sessions.
Period: Overall Study
Arm/Group | TGNC Cohort | Healthcare Participants
Started | 20 | 29
Completed | 14 | 26
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Did not complete pre test or post test survey | 4 | 3

BASELINE CHARACTERISTICS:
Population: Study conducted with transgender and gender non-conforming individuals so gender categories reflect the ways that participants identify.
Groups:
- Total: Total of all reporting groups
Arm/Group | TGNC Cohort | Healthcare Participants | Total
Number analyzed (Participants) | 20 | 29 | 49
Age, Continuous [Mean (Full Range); unit: years] | 27.82 [20 to 77] | 37.65 [24 to 57] | 32.74 [20 to 77]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transwoman/female | 10 | 24 | 34
  Transmen/male | 6 | 3 | 9
  Non-binary/unlabeled | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 29 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 10 | 22 | 32
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 29 | 49
Total Number of Locations to Receive Medical Care Known by TGNC participants [Mean (Full Range); unit: locations] — TGNC participants were asked to name all the locations where they are able to receive care in the Cleveland area. Main hospital systems, specific otherwise -unaffiliated centers and categories were counted. At baseline and post-intervention in a free text field on a survey. Results are only for TGNC participants who completed both pre and post findings Population: Only TGNC participants were asked this question.
  locations
    number analyzed (Participants) | 14 | 0 | 14
    (all) | 3.36 [0 to 11] |  | 3.35 [0 to 11]
Knowledge of transgender and gender nonconforming medical issues [Count of Participants; unit: Participants] — Pre- and post-intervention surveys were completed by participants with questions developed specifically for this study. Participants were asked to respond with their agreement with the following statements: "I know about medical issues that affect transgender and gender nonconforming patients" for Healthcare participants and "I am knowledgeable about how being transgender or gender non-conforming impacts my health" for TGNC participants. Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly.
  Participants
    Strongly Disagree | 0 | 0 | 0
    Disagree | 4 | 7 | 11
    Neutral | 1 | 4 | 5
    Agree | 7 | 11 | 18
    Strongly Agree | 7 | 4 | 11
    No response | 1 | 3 | 4
Ability to Navigate Healthcare System [Count of Participants; unit: Participants] — Pre- and post-intervention surveys were completed by participants with questions developed specifically for this study. TGNC participants were asked " I am able to navigate the healthcare system easily." Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly. Population: This question was only applicable to TGNC participants.
  Participants
    number analyzed (Participants) | 20 | 0 | 20
    Strongly Disagree | 0 |  | 0
    Disagree | 4 |  | 4
    Neutral | 6 |  | 6
    Agree | 5 |  | 5
    Strongly Agree | 3 |  | 3
    No response | 2 |  | 2
Knowledge of How to Express Health and Well-being Concerns [Count of Participants; unit: Participants] — Pre- and post-intervention surveys were completed by participants with questions developed specifically for this study. TGNC participants were asked "I know how to express my concerns about my health and well-being to healthcare providers." Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly. Population: This question was only applicable to TGNC participants.
  Participants
    number analyzed (Participants) | 20 | 0 | 20
    Disagree Strongly | 0 |  | 0
    Disagree | 2 |  | 2
    Neutral | 3 |  | 3
    Agree | 8 |  | 8
    Agree Strongly | 6 |  | 6
    No Response | 1 |  | 1
Comfort in Advocating for Respectful and Appropriate Healthcare [Count of Participants; unit: Participants] — Pre- and post-intervention surveys were completed by participants with questions developed specifically for this study. Healthcare participants were asked "I am comfortable advocating for transgender and gender non-conforming people's right to access respectful and appropriate health care in the place where I practice." Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly. Population: The question was only applicable to Healthcare participants.
  Participants
    number analyzed (Participants) | 0 | 29 | 29
    Disagree Strongly |  | 0 | 0
    Disagree |  | 2 | 2
    Neutral |  | 6 | 6
    Agree |  | 10 | 10
    Agree Strongly |  | 11 | 11
    No Response |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge of TGNC Individuals of Total Number of Locations to Receive Medical Care in Cleveland Known
Description: TGNC participants were asked pre and post-intervention to name all the hospitals they knew of where they could received medical care. Mean and range are reported. This measure was unreliable as participants, when asked in the post survey to name locations for healthcare, were not given those they had identified in the pre-intervention survey, so some participants actually decreased the number they named. Additionally, growth from this measure is mean growth of the group, not a mean of the sum of individual's growth.
Time Frame: Baseline and 11 months
Population: Only TGNC participants who completed pre and post intervention surveys were included.
Measure: Mean (Full Range); unit: locations
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 14 | 0
locations | 3.79 [1 to 13] |

2. Primary Outcome: Change From Baseline in Knowledge of TGNC Cohort About Transgender and Gender Nonconforming Medical Issues
Description: TGNC Cohort Participants were asked to respond with their agreement with the following statement: "I am knowledgeable about how being transgender or gender non-conforming impacts my health." Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly. Change was measured as month 11 minus baseline score, and higher scores represented the better outcome.
Time Frame: Baseline and 11 months
Population: Both the TGNC Cohort and the Healthcare Participant change from baseline in knowledge was measured using the similar question and same scale. TGNC cohort measurement occurred at the first and last date of the TGNC led advocacy meetings (baseline and 11 months later) and the Healthcare Participants measurement occurred at the start and end of their facilitated dialogue with the TGNC Cohort (one 2 hour intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 14 | 0
Participants
  Disagree Strongly | 1 | 0
  Disagree | 1 | 0
  Neutral | 6 | 0
  Agree | 2 | 0
  Agree Strongly | 4 | 0

3. Primary Outcome: Change From Baseline in Knowledge of Healthcare Participants About Transgender and Gender Nonconforming Medical Issues
Description: Healthcare Participants were asked to respond with their agreement with the following statement: "I know about medical issues that affect transgender and gender nonconforming patients." Response options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly. Because healthcare providers only participated in one facilitated dialogue, baseline was measured prior to the dialogue, and post measures were administered the day after the dialogue. Change was measured as post score- baseline score, and higher scores represented the better outcome.
Time Frame: Baseline and 24 hours
Population: The Healthcare Participants measurement occurred at the start and within 24 hours after the end of their facilitated dialogue with the TGNC Cohort (one 2 hour intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 0 | 26
Participants
  Disagree Strongly | 0 | 0
  Disagree | 0 | 2
  Neutral | 0 | 3
  Agree | 0 | 15
  Agree Strongly | 0 | 6

4. Primary Outcome: Change From Baseline in Attitude of TGNC Individuals Towards Navigating Their Interactions With Healthcare Providers.
Description: TGNC Individuals were asked to respond with their agreement with the following two statements:
  1. "I am able to navigate the healthcare system easily", and
  2. "I know how to express my concerns about my health and well-being to healthcare providers." Response options were 1=Disagree Strongly, 2-=Disagree, 3=Neutral, 4=Agree and 5=Strongly agree. For these questions, a higher score indicated confident attitude in handling their healthcare needs. Change from Baseline to 11 months was measured.
Time Frame: Baseline and 11 months
Population: Only the TGNC (n=14) were asked these questions at baseline (pre-intervention) and 11 months (post-intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 14 | 0
Participants
  I am able to navigate the healthcare system easily: Disagree Strongly | 0 |
  I am able to navigate the healthcare system easily: Disagree | 3 |
  I am able to navigate the healthcare system easily: Neutral | 1 |
  I am able to navigate the healthcare system easily: Agree | 6 |
  I am able to navigate the healthcare system easily: Agree Strongly | 4 |
  I am able to navigate the healthcare system easily: No response | 0 |
  I know how to express my concerns about my health and well-being to healthcare providers.: Disagree Strongly | 0 |
  I know how to express my concerns about my health and well-being to healthcare providers.: Disagree | 1 |
  I know how to express my concerns about my health and well-being to healthcare providers.: Neutral | 5 |
  I know how to express my concerns about my health and well-being to healthcare providers.: Agree | 2 |
  I know how to express my concerns about my health and well-being to healthcare providers.: Agree Strongly | 6 |
  I know how to express my concerns about my health and well-being to healthcare providers.: No response | 0 |

5. Primary Outcome: Change in Attitude of Medical Providers Towards Transgender Issues.
Description: Healthcare Participants were asked to respond with their agreement with the following statement: "I am comfortable advocating for transgender and gender non-conforming people's right to access respectful and appropriate health care in the place where I practice." Response Options were 1=Disagree Strongly, 2=Disagree, 3=Neutral, 4=Agree, and 5=Agree Strongly, with a higher score indicating a more positive attitude towards transgender issues. Change was measured by subtracting the providers' responses after participation in a facilitated dialogue with TGNC participants from their scored response prior to participating in the dialogue.
Time Frame: Baseline and 24 hours.
Population: Only Healthcare Participants were asked this question.
Measure: Count of Participants; unit: Participants
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 0 | 26
Participants
  Disagree Strongly |  | 0
  Disagree |  | 1
  Neutral |  | 1
  Agree |  | 10
  Agree Strongly |  | 14
  No response |  | 0

6. Primary Outcome: Qualitative Shift in Confidence of TGNC Individuals in Seeking Medical Care After the Intervention.
Description: Percentage of TGNC individuals expressing key themes related to shift of confidence of TGNC Individuals to seek medical care following the intervention.
Time Frame: Interview at 11 months.
Population: Amongst the 8 TGNC participants who agreed to be interviewed following the intervention, a key theme in the qualitative evaluation was a sense of personal growth in confidence regarding speaking up both inside and outside of healthcare settings.
Measure: Count of Participants; unit: Participants
Arm/Group | TGNC Cohort | Healthcare Participants
Number analyzed (Participants) | 8 | 0
Participants | 8 | 0

7. Primary Outcome: Qualitative Shift in Confidence of Medical Provider in Providing Culturally Competent Medical Care to TGNC Individuals After the Intervention.
Description: The number of medical providers expressing themes illustrating a shift in confidence with their ability to provide culturally competent medical care in structured interview following the facilitated dialogue with members of the TGNC participant group.
Time Frame: Interview within one day following the facilitated dialogue
Population: This was a qualitative interview and analysis was for only the 8 healthcare participants who agreed to the structured interviews following the intervention in structured interviews.
Measure: Number; unit: percentage of hc participants
Arm/Group | Healthcare Participants
Number analyzed (Participants) | 8
percentage of hc participants
  Expressing confidence in structured interview | 6
  Expressing no confidence in structured interview: number analyzed (Participants) | 2
  Expressing no confidence in structured interview | 2

ADVERSE EVENTS:
Time Frame: 22 months following the participants' first meeting of the study.
Groups:
- Healthcare Participants: Healthcare providers and staff who attended a facilitated dialogue with TGNC Cohort to address barriers to access and to enter into dialogue with Transgender and gender non-conforming (TGNC) identifying individuals.
Arm/Group | TGNC Cohort | Healthcare Participants
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/29
Other Adverse Events (participants affected / at risk) | 0/20 | 0/29

LIMITATIONS AND CAVEATS:
The Translate Study was a pilot study, with a convenience sampling design that limits the findings' generalizability. Sample size and inability to use a validated scale limits the findings' reliability. The surveys were developed before assembling the TGNC cohort so the questions did not always align with their objectives. One healthcare participant complained that the facilitated dialogue with TGNC cohort unnecessarily discussed racism.

The Study PI and staff are no longer employed by CWRU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03808883/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03808883/ICF_001.pdf